CLINICAL TRIAL: NCT06829836
Title: Can You Breathe Your Way To Better Health?
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Northern Colorado (Other)
Responsible Party: Principal Investigator, Laura Stewart, Professor, University of Northern Colorado
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2404058931
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Chronic Stress; Autonomic Dysfunction
Keywords: High intensity interval training (HIIT); Cyclic hyperventilation with retention (CHR); intervention; Natural killer cells; training; stress; autonomic nervous system; innate immune system; natural killer cell cytotoxicity; heart rate variability (HRV)
MeSH Terms: conditions — Neoplasms; Primary Dysautonomias | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CON, control (No Intervention): The control group will undergo the same testing procedures outlined above, but they will be asked to maintain their current level of activity and normal daily habits for the duration of the intervention.
- HIG, High intensity group (Active Comparator): During the exercise session, HR will be measured via a Polar heart rate strap (Kempele, Finland). The training sessions will consist of six 90-second high-intensity cycling (HIC) sprints performed on a cycle ergometer (Monark Ergomedic 895E, Monark, Varberg, Sweden) at 80-90% VO2max, followed by 180 seconds of low-intensity cycling (LIC) at 50-60% of VO2max. During both HIC and LIC intensities, participants will be asked rate of perceived exertion, which will be compared to the participants' heart rate throughout the exercise sessions. This supervised training protocol will require 9 minutes of HIC at 80-90% VO2max and 18 minutes of LIC at 50-60% VO2max. The cycling session will begin with a brief warm-up and end with a cool-down down totaling the entire supervised exercise session for 30 minutes. Training sessions will be performed 48 hours after the previous training session for a total of 3 times per week on Mondays, Wednesdays, and Fridays.
  Interventions: Behavioral: Hight intensity interval training
- CHG, Cyclic hyperventilation group (Active Comparator): The breathing intervention will consist of a daily breathing practice lasting 5 to 10 minutes for 5 days per week. Breathing practice is a form of cyclic hyperventilation consisting of 30 breath (inhalation and exhalation) repetitions followed by an exhaled breath retention for 15 seconds during the first week and up to 30 seconds during the second week. A total of 3 rounds will be performed by the participants. Participants will be instructed to perform breathing repetitions in a controlled and consistent manner while either seated or lying down. Participants will receive guided instruction via a video on breath cycle queues, informing the participants when to inhale, exhale, and when to retain their breath while being supervised by the research team via Zoom call. Upon completion of the breath training sessions, the research team will conduct a guided cooldown and check in with all participants to ensure they are feeling no adverse side effects from the breathing exercise.
  Interventions: Behavioral: Cyclic Hyperventilation with Retention

INTERVENTIONS:
Behavioral: Hight intensity interval training — Participants assigned to this intervention group will complete 6 supervised HIIT sessions over 2 weeks.
  Other Names: HIIT; SIT; Sprint interval training
  Arms: HIG, High intensity group
Behavioral: Cyclic Hyperventilation with Retention — Participants of this intervention group will complete a total of 10 remote guided breathing sessions on Zoom over 2 weeks.
  Other Names: CHR
  Arms: CHG, Cyclic hyperventilation group

SUMMARY:
The purpose of this clinical trial is to explore the effects of either a 2-week high-intensity interval training (HIIT) or breath training intervention on measures of overall health, circulating biomarkers of stress, and immune function.

Specific aims include: - Does a 2-week HIIT or breath training intervention improve measurements of overall health, including heart rate variability, physical activity, sleep quality, and severity of depression, anxiety, and stress? -Does a 2-week HIIT or breath training intervention improve circulating concentrations of stress-related biomarkers? Does a 2-week HIIT or breath training intervention improve immune function? Researchers will compare HIIT and breath training to see if equivalent immune improvements are observed.

Participants will: -Undergo 2 weeks of HIIT or breath training interventions at a frequency of 3 times per week for 30 minutes or 5 times per week for 5 minutes if placed into an intervention group. -Undergo testing measures at the two pre- and post-intervention time points, if placed in the intervention groups or the healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* Age, 18-50 years
* Sex, Male and Female
* Informed Consent, The capability and willingness to give written informed consent to understand the exclusion criteria and to accept the randomized group assignment is required.
* PAR-Q+, The capability and willingness to complete the physical activity readiness questionnaire, with no medical clearance needed.
* Physical Activity: Participants must refrain from regular HIIT and structured breathing practices for a month before participation
* Depression, Anxiety, and Stress Scale, Subcategory Scoring (DASS-21) Participants must score in the mild or greater category for Depression, Anxiety, and Stress. Depression ≥ 10, Anxiety ≥ 8, and Stress ≥ 14.

Exclusion Criteria:

* Age: Individuals under 18 years and over 50 years
* Significant Respiratory Conditions, including but not limited to asthma, chronic obstructive pulmonary disease,
* Significant Cardiovascular Disease: Participants with a known cardiovascular condition such as a previous myocardial infarction, congestive heart failure, stroke, or transient ischemic attack, cardiomyopathy, serious arrhythmia, peripheral vascular disease, untreated atherosclerosis, or hypertension.
* Significant Musculoskeletal Disease, including but not limited to osteopenia, osteoporosis, rheumatoid arthritis, and sarcopenia
* Cognitive and Mental Health, including but not limited to untreated anxiety, untreated depression, post-traumatic stress disorder, and thoughts of suicide.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Serum Analysis: C-reactive protein (CRP) | Visit 1(Week 1) and Visit 3 (Week 4): 15 minutes for blood draw. The assay itself takes 3 hours.
  Approximately 60 mL of whole blood will be collected into serum separator tubes (Beckton Dickinson, East Rutherford, NJ, USA), allowed to clot for 30-min at room temperature, and then centrifuged at 2000 RPM for 15 min. The serum will be pipetted into 1.5 mL microcentrifuge tubes (Eppendorf AG, Hamburg, Germany) and immediately stored in a -80 °C freezer. Serum concentrations of CRP will be determined with a commercially available enzyme-linked immunosorbent assay (ALPCO Diagnostics, Salem, NH, USA). Microplates will be read with an ELx800 BioTek microplate reader (BioTek Instruments, Inc., Winooski, VT, USA) at the recommended wavelength of 450 nanometers.
Serum Analysis: Brain Derived Neurotrophic Factor (BDNF) | Visit 1A (Week 1) and Visit 2A (Week 4): 15 minutes for blood draw. The assay itself takes 3 hours.
  Approximately 40 mL of whole blood will be collected into serum separator tubes (Beckton Dickinson, East Rutherford, NJ, USA), allowed to clot for 30 minutes at room temperature, and then centrifuged at 2000 RPM for 15 min. The serum will be pipetted into 1.5 mL microcentrifuge tubes (Eppendorf AG, Hamburg, Germany) and immediately stored in a -80 °C freezer. Serum concentrations of BDNF (Sigma-Aldrich, St. Louis, MO, USA) will be determined with commercially available enzyme-linked immunosorbent assays. Microplates will be read with an ELx800 BioTek microplate reader (BioTek Instruments, Inc., Winooski, VT, USA) at the recommended wavelength of 450 nanometers.
Natural Killer cell quantity | Visit 1(Week 1) and Visit 3 (Week 4): 15 minutes for blood draw. The assay itself takes ~10-12 hours.
  15mL of whole blood will be obtained using sodium heparin tubes and a peripheral venous puncture. Blood samples will be mixed with Dulbecco's phosphate buffer solution (DPBS) at a 1:1 ratio and layered over 20 mL of Ficoll gradient matrix. Blood samples will be centrifugation at 111 x g for 40 minutes, acceleration 7, brake 0 (Eppendorf 5810R centrifuge, Hamburg, Germany). Samples will be washed 3 times, then resuspended at 1.0 * 10^6 cells/mL and incubated for 4 hours at 37 degrees Celsius, with 5% CO2. Next, samples will be pelleted, resuspended, and antibody-receiving samples will each receive 500uL DPBS and 1uL of Fragment crystabillize blocker (FcB)/1.0*10^6 cells and incubate on ice for 20 minutes. Samples will be pelleted, resuspended in 500uL DPBS and receive 500uL of DPBS and 2uL of CD56 (NCAM) monoclonal antibodies, incubate on ice for 20 minutes, pelleted, and resuspended in 1mL of DPBS, then analyzed using an Attune NXT flow cytometer (Thermo Fischer, Waltham, MA).
Natural Killer Cell Cytotoxicity | Visit 1(Week 1) and Visit 3 (Week 4): 15 minutes for blood draw. The assay itself takes ~10-12 hours.
  Chronic human myelogenous leukemia cells (K562; ATCC, Manassas, VA) are used to evaluate NKC effector function. K562 cells are stained with Alexa-Fluor 647-conjugated anti-CD71. K562 cells are further stained with Calcein-AM viability dye (Thermo Fisher Scientific, Waltham, MA), then incubated on ice for 20 min. K562 cells are washed and resuspended at 1.0 × 106 cells/mL in complete RPMI 1640 medium. Human PBMCs containing effector NK and NKT cells are co-cultured with K562 cells in 5 mL Eppendorf tubes at a 40:1 PBMC: K562 effector: target (E: T) ratio and incubated for 4 h at 37 °C in a cell incubator. Following co-incubation, samples are centrifuged at 400 x g for 5 min and resuspended in ice-cold DPBS for analysis. After the 4-hour co-culture, these samples are analyzed via flow cytometry to determine the total proportion of alive (Calcein-AM+/CD71+) versus estimated K562 cells. Changes in proportion and MFI of these populations were further analyzed using Floreada.io.
Heart Rate Variability (HRV) | Visit 2 (week 1) and Vist 4 (week 4)
  Heart rate variability (HRV) will be analyzed to determine the fluctuation in the time intervals between adjacent heartbeats to assess autonomic regulation of the heart. Resting HR and HRV were measured using the electrocardiograph (GE CASE Exercise Testing System Version 6.0, Chicago, Illinois). To measure HRV, the standard deviation of normal to normal beats (SDNN) was used with the 10-second electrocardiogram reading. Based on the outcome of this assessment, participants with SDNN values below 50 ms will be classified as unhealthy, 50-100 ms will be classified as having compromised health, and above 100 ms will be classified as healthy.

SECONDARY OUTCOMES:
Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) | Visit 1 (week 1) 10 minutes
  PAR-Q+ utilizes yes or no generalized health questions to screen participants interested in engaging in an exercise program for the need of medical clearance and physician release. The PAR-Q+ has 7 general health questions ranging from Does the participant feel chest pain at rest or during activities of daily living? Individuals who are eligible for this investigation require no further medical clearance before participating in an exercise program and should truthfully answer NO to every question. Participants who answer "Yes" to any questions will be required to answer follow-up questions to determine the need for medical clearance. If medical clearance is suggested, the individual will not be eligible to participate.
Depression Anxiety and Stress Scale (DASS-21) | Visit 1 (week 1) and Visit 3 (week 4) 10 minutes each
  The DASS-21 contains 3 subscales assessing Depression, Anxiety, and Stress consisting of 7 questions for each subscale, where a high score of 28+ indicates "Extremely Severe" levels of Depression, a high score of 20+ indicates "Extremely Severe" levels of Anxiety, and a high score of 34+ indicates "Extremely Severe" levels of Stress, while low scores of 0-9 indicates "Normal" levels of Depression, scores of 0-7 indicates "Normal" levels of Anxiety, and scores of 0-14 indicates "Normal" levels of Stress. Raw scores for each subcategory will be recorded and multiplied by 2 to calculate the subcategory score.
Pittsburg Sleep Quality Index (PSQI) | Visit 1 (week 1) and Visit 3 (week 4) 10 minutes each
  Participants will be asked to complete a paper version of the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a 19-question self-reported sleep quality tool divided into 7 subcategories for scoring: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Five additional questions directed to the respondent's roommate or bed partner are not used in the scoring but are utilized for clinical purposes.
Wisconsin Upper Respiratory Symptom Survey (WURSS-21) | Visit 1 (week 1) and Visit 3 (week 4) 10 minutes each
  The WURSS is an illness-specific quality of life measurement designed to assess the impact of the common cold (acute upper respiratory infection). It consists of 21 questions that investigate the perception of sickness, the severity of sickness-related symptoms over the last 24 hours, the extent to which sickness has hindered the ability to think clearly and accomplish daily tasks over the past 24 hours, and the comparison of sickness to the day before.
Physical Activity and Sleep Tracking | 4 weeks
  Heart rate, sleep duration, and steps will be measured and obtained via the WHOOP Strap 4. Measures obtained from the WHOOP strap include continuous heart rate monitoring, sleep cycle, sleep stage, and total step data. The HRV measurement from the WHOOP strap will then be compared to the HRV analysis performed using the standard deviation of the normal-to-normal beat method.
VO2Max | Visit 2 (week 1) 30-45 minutes
  Maximal oxygen consumption will be assessed on a cycle ergometer using a TrueOne 2400 Metabolic Measurement System. A Polar Heart Rate Sensor H1 will be outfitted for each participant before starting the assessment. Participants will rest for 5 minutes in a seated position when heart rate, blood pressure, and blood lactate are measured. Next, the participant will be fitted to the cycle ergometer and perform a brief 5-minute warm-up at 0.5 kg and 60 rpm. Next, the pedal cadence increases to 75-85 rpm, and the participant starts stage 1. Every stage lasts 3 minutes, at the end of every stage, heart rate, blood lactate, blood pressure, and RPE are recorded, and 0.5 kg of resistance is added to the weight basket. Once blood lactate concentration is above 4.0 mmol/L, an incremental increase of 0.2 kg occurs. Assessment is terminated after volitional fatigue, failure to maintain pedal cadence, failure to increase heart rate or VO2 in subsequent stages, and the participant's request.

OTHER OUTCOMES:
Anthropometric Measures: Height | Visit 1 (week 1)
  Height will be obtained in centimeters (cm)( using a stadiometer SECA 220 (Chino, California, USA).
Anthropometric Measures: Weight | Visit 1 (week 1)
  Weight will be obtained in kilograms (kg) using a Detecto standing digital scale (Webb City, Missouri, USA).
Anthropometric Measures: Lean Body Mass | Visit 1 (week 1)
  Lean body mass (LBM) will be measured in kilograms and evaluated using air displacement plethysmography using a calibrated BOD POD (COSMED USA Inc., Concord, CA).
Anthropometric Measures: Body Fat Percentage | Visit 1 (week 1)
  Body fat percentage (BF%) will be measured as a percentage of estimated body fat relative to total body mass and evaluated using air displacement plethysmography using a calibrated BOD POD (COSMED USA Inc., Concord, CA).
Hydration | Visit 1, Visit 2 (week 1) and Visit 3 (Week 4)
  A refractometer (Atago, Tokyo, JPN) will be used to evaluate urine-specific gravity with a dehydration cutoff point set to ≥1.020 mg/dL. Dehydrated participants will be given time to hydrate. If dehydration persists, participants will be asked to reschedule the session. After verbal compliance and hydration status are confirmed, participants will proceed with the study's procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Northern Colorado, 1610 Gunter Hall, 1828 10th Ave, Greeley, CO 80631, Greeley, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make all study documents available by reasonable request (Laura.stewart@unco.edu) up to 3 years after data collection is complete.
Time Frame: Start: Jan 27, 2025 - Jan 27, 2028
Access Criteria: Anyone who contacts Laura.stewart@unco.edu with a reasonable request.